CLINICAL TRIAL: NCT02178410
Title: Vitamin D and Omega-3 Trial (VITAL Rhythm Study)
Brief Title: VITAL Rhythm Study
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Christine M. Albert, MD, MPH, Principle Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012P002146; R01HL116690 (NIH)
Record Dates: First submitted 2014-06-25; First posted 2014-06-30 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Disease
Keywords: Atrial Fibrillation; Vitamin D3; Omega-3 fatty acids; Fish oil
MeSH Terms: conditions — Cardiovascular Diseases; Atrial Fibrillation | interventions — Cholecalciferol; Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (4):
- Vitamin D + fish oil (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D3; Drug: Omega-3 fatty acids (fish oil)
- Vitamin D + fish oil placebo (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Fish oil placebo
- Vitamin D placebo + fish oil (Active Comparator)
  Interventions: Drug: Omega-3 fatty acids (fish oil); Dietary Supplement: Vitamin D3 placebo
- Vitamin D placebo + fish oil placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Fish oil placebo; Dietary Supplement: Vitamin D3 placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 (cholecalciferol), 2000 IU per day.
  Other Names: cholecalciferol
  Arms: Vitamin D + fish oil; Vitamin D + fish oil placebo
Drug: Omega-3 fatty acids (fish oil) — Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Arms: Vitamin D + fish oil; Vitamin D placebo + fish oil
Dietary Supplement: Fish oil placebo — Fish oil placebo
  Arms: Vitamin D + fish oil placebo; Vitamin D placebo + fish oil placebo
Dietary Supplement: Vitamin D3 placebo — Vitamin D3 placebo
  Arms: Vitamin D placebo + fish oil; Vitamin D placebo + fish oil placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL) is an ongoing randomized clinical trial of 25,871 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor® fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in individuals who do not have a prior history of these illnesses. The purpose of this ancillary study is to ascertain and adjudicate atrial fibrillation (AF) outcomes for the primary aim of testing whether omega-3 fatty acid and/or vitamin D supplementation influence atrial fibrillation risk in the general population. We also plan to examine how these agents might impact the development of AF subtypes (persistent versus paroxysmal), intermediate phenotypes for heart rhythm disorders (electrocardiographic parameters), as well as explore effects on arrhythmic death and whether baseline blood levels and/or race modify treatment effects.

DETAILED DESCRIPTION:
Atrial fibrillation and sudden cardiac death assessments, as well as blood analyses, will be conducted on the entire VITAL Study population, and ECG analyses will be limited to the Clinical and Translational Science Center (CTSC) sub-cohort of 1,054 VITAL participants who live near the Boston area and agree to participate in a series of ancillary studies in addition to the main trial.

Investigators will ascertain atrial fibrillation events utilizing self-report of physician diagnoses of atrial fibrillation received on annual questionnaires from study participants supplemented by outpatient and hospital visits for AF identified through Centers for Medicare and Medicaid Services (CMS) data linkage. Investigators will also ascertain additional information regarding atrial fibrillation diagnosis from supplementary questionnaires, and seek consent to review all inpatient and outpatient hospital records pertaining to atrial fibrillation diagnosis and evaluation. Atrial fibrillation events will be confirmed by an endpoint committee composed of cardiologists, which will also make a determination on atrial fibrillation subtype and pattern. Questionnaires that inquire about recurrent atrial fibrillation events, pattern of AF, latest medical record evaluation and treatments for AF will be sent to participants with confirmed atrial fibrillation. Medical records will be requested and reviewed an endpoint committee to determine atrial fibrillation subtype and progression. An intention-to-treat analysis examining the 5-year treatment effects of omega-3 fatty acids and vitamin D on incident atrial fibrillation, as well as subtypes at the time of diagnosis will be performed to address the primary aims. We will repeat these analyses at the end of extended follow-up to assess cumulative and post-treatment effects of omega-3 fatty acids and vitamin D and AF subtypes two years after diagnosis.

Electrocardiograms will be obtained at baseline and again after two years of treatment and follow-up among a sub-cohort of 1,054 patients being enrolled in VITAL at the CTSC. Investigators will utilize these ECG data to evaluate whether treatment with omega-3 fatty acids and vitamin D3 have significant effects on ECG measures. The ECGs will also be utilized to estimate the prevalence of asymptomatic persistent atrial fibrillation in our population not detected by our atrial fibrillation surveillance methods.

Investigators will examine baseline blood samples for participants with confirmed atrial fibrillation for the purpose of exploring whether the effect of vitamin D3 or fish oil supplementation on atrial fibrillation risk varies by the baseline blood levels of these nutrients.

Investigators will also seek additional information necessary to classify deaths as sudden or arrhythmic in origin, and cardiac deaths will be reviewed by an endpoint committee of cardiologists. Once these results have been compiled investigators will explore whether omega-3 fatty acids and/or vitamin D might have an effect on sudden and/or arrhythmic cardiac death.

ELIGIBILITY:
To be eligible this ancillary study participants must be enrolled in the Vitamin D and Omega-3 Trial (VITAL; National Clinical Trial (NCT) 01169259) and meet the following criteria:

Inclusion Criteria:

- physician diagnosis of atrial fibrillation after randomization

and/or

- cardiovascular death

Exclusion Criteria:

- physician diagnosis of atrial fibrillation prior to randomization

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25119 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Atrial Fibrillation | 7 years
  To assess whether omega-3 fatty acids (Omacor® 840 mg eicosapentaenoic acid (EPA) + docosahexaenoic acid (DHA) or vitamin D3 supplementation influences risk of atrial fibrillation in a general population of men and women without prior cardiovascular disease.

SECONDARY OUTCOMES:
Atrial Fibrillation | 7 years
  To examine the short and long-term impacts of vitamin D3 and EPA+DHA supplementation on the development of AF subtypes.
Arrhythmic endpoints | 5 years
  To examine the effect of vitamin D3 or EPA+DHA supplementation on electrocardiographic parameters to further understand mechanisms underlying associations with arrhythmic endpoints.

OTHER OUTCOMES:
Sudden Cardiac Death | 5 years
  To explore effects of arrhythmic death and whether baseline blood levels and/or race modify treatment effects.

CONTACTS AND LOCATIONS:
Overall Officials: Christine M. Albert, M.D., M.P.H., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Qian F, Tintle N, Jensen PN, Lemaitre RN, Imamura F, Feldreich TR, Nomura SO, Guan W, Laguzzi F, Kim E, Virtanen JK, Steur M, Bork CS, Hirakawa Y, O'Donoghue ML, Sala-Vila A, Ardisson Korat AV, Sun Q, Rimm EB, Psaty BM, Heckbert SR, Forouhi NG, Wareham NJ, Marklund M, Riserus U, Lind L, Arnlov J, Garg P, Tsai MY, Pankow J, Misialek JR, Gigante B, Leander K, Pester JA, Albert CM, Kavousi M, Ikram A, Voortman T, Schmidt EB, Ninomiya T, Morrow DA, Bayes-Genis A, O'Keefe JH, Ong KL, Wu JHY, Mozaffarian D, Harris WS, Siscovick DS; Fatty Acids and Outcomes Research Consortium (FORCE). Omega-3 Fatty Acid Biomarkers and Incident Atrial Fibrillation. J Am Coll Cardiol. 2023 Jul 25;82(4):336-349. doi: 10.1016/j.jacc.2023.05.024. PMID 37468189
- [Result] Gencer B, Djousse L, Al-Ramady OT, Cook NR, Manson JE, Albert CM. Effect of Long-Term Marine ɷ-3 Fatty Acids Supplementation on the Risk of Atrial Fibrillation in Randomized Controlled Trials of Cardiovascular Outcomes: A Systematic Review and Meta-Analysis. Circulation. 2021 Dec 21;144(25):1981-1990. doi: 10.1161/CIRCULATIONAHA.121.055654. Epub 2021 Oct 6. PMID 34612056
- [Result] Middeldorp ME, Sandhu RK, Mao J, Gencer B, Danik JS, Moorthy V, Cook NR, Albert CM. Risk Factors for the Development of New-Onset Persistent Atrial Fibrillation: Subanalysis of the VITAL Study. Circ Arrhythm Electrophysiol. 2023 Dec;16(12):651-662. doi: 10.1161/CIRCEP.123.012334. Epub 2023 Nov 29. PMID 38018439
- [Result] Siddiqi HK, Vinayagamoorthy M, Gencer B, Ng C, Pester J, Cook NR, Lee IM, Buring J, Manson JE, Albert CM. Sex Differences in Atrial Fibrillation Risk: The VITAL Rhythm Study. JAMA Cardiol. 2022 Oct 1;7(10):1027-1035. doi: 10.1001/jamacardio.2022.2825. PMID 36044209
- [Result] Albert CM, Cook NR, Pester J, Moorthy MV, Ridge C, Danik JS, Gencer B, Siddiqi HK, Ng C, Gibson H, Mora S, Buring JE, Manson JE. Effect of Marine Omega-3 Fatty Acid and Vitamin D Supplementation on Incident Atrial Fibrillation: A Randomized Clinical Trial. JAMA. 2021 Mar 16;325(11):1061-1073. doi: 10.1001/jama.2021.1489. PMID 33724323
- [Derived] Tikkanen JT, Soliman EZ, Pester J, Danik JS, Gomelskya N, Copeland T, Lee IM, Buring JE, Manson JE, Cook NR, Albert CM. A randomized clinical trial of omega-3 fatty acid and vitamin D supplementation on electrocardiographic risk profiles. Sci Rep. 2023 Jul 15;13(1):11454. doi: 10.1038/s41598-023-38344-x. PMID 37454148
- See also: Welcome to the VITAL Study website — http://www.vitalstudy.org/